CLINICAL TRIAL: NCT02975609
Title: Phase II Trial of Stereotactic Body Radiation Therapy Compared With Conventional Fractionated Radiotherapy for Oligometastatic Non-Small Cell Lung Cancer
Brief Title: Phase II Trial of SBRT Compared With Conventional Radiotherapy for Oligometastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Director, Department of Radiation Oncology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHLC008
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: NSCLC
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Fractionated Radiotherapy (Active Comparator): The patients enrolled receive firstly 4-6 cycles chemotherapy (platinum-based doublet chemotherapy), and achieve response(stable disease or partial response or complete response). Patients will be randomized into the control group undergoing the conventional fractionated radiotherapy to all metastatic sites and the primary tumor.
  Interventions: Radiation: Conventional Fractionated Radiotherapy
- Stereotactic Body Radiation Therapy (Experimental): The patients enrolled receive firstly 4-6 cycles chemotherapy (platinum-based doublet chemotherapy), and achieve response(stable disease or partial response or complete response). Patients will be randomized into the experimental group undergoing SBRT to all metastatic sites and the primary tumor.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Conventional Fractionated Radiotherapy — 5Fx/W,3Gy/Fx,Dt:PTV-G:30Gy/10F/2W for metastatic sites, Dt:60Gy/30F for primary tumor and metastatic lymph node.
  Arms: Conventional Fractionated Radiotherapy
Radiation: Stereotactic Body Radiation Therapy — 30Gy/3-5F for the primary and the metastases.
  Arms: Stereotactic Body Radiation Therapy

SUMMARY:
This protocol is a phase II randomized controlled trial (RCT) evaluating the efficacy of SBRT compared with conventional fractionated radiotherapy for oligometastatic Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
Non small-cell lung cancer (NSCLC) is the leading cause of cancer-related death worldwide. Approximately half of all patients with NSCLC present with metastatic disease at the time of diagnosis, and the predominant pattern of failure in patients with localized NSCLC is distant metastatic spread. The standard treatment in metastatic disease is cytotoxic chemotherapy with a mean overall survival between 8-11 months.

Various studies suggest that patients who clinically present with a limited number of metastases, a term defined as oligometastatic disease, could have a better prognosis of survival with a radical treatment, than for their counterparts with a greater number of metastasis. Much of the current clinical outcomes in oligometastatic disease is based on a series of the retrospective studies.

This is a randomised prospective phase II study based on patients with stage IV oligometastatic NSCLC according to UICC stage system(version 7,2009) or oligometastatic disease after radical operation for stage I-III NSCLC. The purpose of this study is to add more information to the current medical literature about the efficacy and safety of Stereotactic Body Radiation Therapy (SBRT) compared with conventional fractionated radiotherapy for oligometastatic non-small cell lung cancer (equal to or less than 5 sites and equal to or less than 5cm in maximum diameter).

The patients enrolled receive firstly 4-6 cycles chemotherapy (platinum-based doublet chemotherapy), and achieve response(stable disease or partial response or complete response). Patients will be randomized into two groups. The control group will undergo the conventional fractionated radiotherapy to all metastatic sites and the primary tumor. The experimental group will receive SBRT to primary lesions or metastatic lesions.

The investigators will compare progress free survival(PFS) ,overall survival, incidence of treatment-related adverse events of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small-cell lung cancer.
* Stage IV oligometastatic NSCLC according to UICC stage system(version 7,2009) or oligometastatic disease after radical operation for stage I-III NSCLC.
* The patients receive firstly 4-6 cycles chemotherapy (platinum-based doublet chemotherapy), and achieve response(stable disease or partial response or complete response).
* Staging with chest CT scan, abdominal ultrasonography , MRI brain, Bone scan and/or FDG PET-CT whole body scan.
* Number of metastatic lesions equal to or less than 5.
* Maximum diameter of metastatic tumors equal to or less than 5cm.
* ECOG performance status 0-2 at time of registration.
* EGFR testing is mandatory.
* No brain metastasis in MRI.
* No liver metastasis in abdominal CT or MRI.
* No malignant pleural effusion or pericardial effusion or peritoneal effusion.
* Acceptable lung function for radical lung radiotherapy.
* Stable lab values: Hematological:

Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin≥9 g/dL Renal: Creatinine OR Measured or calculated creatinine clearance (CrCl)(glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5×the upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels>1.5× institutional ULN Hepatic: Total bilirubin ≤1.5×ULN OR Direct bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN,globulin≥20 g/L, albumin≥30 g/L.

* No relevant co-morbidities, including pulmonary fibrosis and connective tissue disorders
* Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

* Patient has had palliative radiotherapy to any tumour site prior to registration and/or requires palliative radiotherapy prior to randomisation.
* Patient has received any molecular targeted therapeutic drugs for NSCLC malignancy.
* The patients receive firstly 4-6 cycles chemotherapy (platinum-based doublet chemotherapy), and achieve progressive disease.
* Any unstable systemic disease, including active infection, uncontrolled high blood pressure, unstable angina, newly observed angina pectoris within the past 3 months, congestive heart failure (New York heart association (NYHA) class II or higher), myocardial infarction onset six months before included into the group, and severe arrhythmia, liver, kidney, or metabolic disease in need of drug therapy.
* Previously diagnosed with immunodeficiency disease.
* Human immunodeficiency virus (HIV) infection.
* Women in pregnancy or lactation.
* Patients with mental illness, considered as "can't fully understand the issues of this research".
* other Cancer history.
* Histologically confirmed small cell carcinoma or other non NSCLC compositions in the cancer tissue.
* Brain metastasis or liver metastasis or malignant pleural effusion or pericardial effusion or peritoneal effusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Incidence of treatment-related adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Fu, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salama JK, Schild SE. Radiation therapy for oligometastatic non-small cell lung cancer. Cancer Metastasis Rev. 2015 Jun;34(2):183-93. doi: 10.1007/s10555-015-9559-z. PMID 25948377
- [Background] Hanna GG, Landau D. Stereotactic body radiotherapy for oligometastatic disease. Clin Oncol (R Coll Radiol). 2015 May;27(5):290-7. doi: 10.1016/j.clon.2015.02.003. Epub 2015 Mar 12. PMID 25770653
- [Background] Tree AC, Khoo VS, Eeles RA, Ahmed M, Dearnaley DP, Hawkins MA, Huddart RA, Nutting CM, Ostler PJ, van As NJ. Stereotactic body radiotherapy for oligometastases. Lancet Oncol. 2013 Jan;14(1):e28-37. doi: 10.1016/S1470-2045(12)70510-7. PMID 23276369
- [Background] Ashworth A, Rodrigues G, Boldt G, Palma D. Is there an oligometastatic state in non-small cell lung cancer? A systematic review of the literature. Lung Cancer. 2013 Nov;82(2):197-203. doi: 10.1016/j.lungcan.2013.07.026. Epub 2013 Aug 20. PMID 24051084
- [Background] Ashworth AB, Senan S, Palma DA, Riquet M, Ahn YC, Ricardi U, Congedo MT, Gomez DR, Wright GM, Melloni G, Milano MT, Sole CV, De Pas TM, Carter DL, Warner AJ, Rodrigues GB. An individual patient data metaanalysis of outcomes and prognostic factors after treatment of oligometastatic non-small-cell lung cancer. Clin Lung Cancer. 2014 Sep;15(5):346-55. doi: 10.1016/j.cllc.2014.04.003. Epub 2014 May 15. PMID 24894943